CLINICAL TRIAL: NCT06678451
Title: Effect of Sugammadex on Quality of Recovery Following Laparoscopic Bariatric Surgery
Brief Title: Sugammadex on Laparoscopic Bariatric Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YXLL-2024-195
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Laparoscopic Bariatric Surgery; Sugammadex
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex group (Experimental): When T2 appeared, the sugammadex group was given 2mg/kg of sugammadex intravenously (adjusted body weight)
  Interventions: Drug: Sugammadex
- Neostigmine group (Active Comparator): When T2 appeared, the neostigmine group was given 0.04mg/kg of neostigmine + 0.02mg/kg of atropine intravenously (adjusted body weight).
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — When T2 appeared, the sugammadex group was given 2mg/kg of sugammadex intravenously (adjusted body weight), the neostigmine group was given 0.04mg/kg of neostigmine + 0.02mg/kg of atropine intravenously (adjusted body weight).
  Arms: Sugammadex group
Drug: Neostigmine — When T2 appeared, the neostigmine group was given 0.04mg/kg of neostigmine + 0.02mg/kg of atropine intravenously (adjusted body weight).
  Arms: Neostigmine group

SUMMARY:
Laparoscopic bariatric surgery has been recognized as the most effective treatment for obesity and related metabolic diseases. Because obesity patients often associated with sleep apnea syndrome or obesity hypoventilation syndrome, combined with the residual effect of muscle relaxants during the operation is easy to lead to respiratory obstruction and respiratory insufficiency, and hypoxemia and carbon dioxide retention are easy to occur after surgery, Post-extubation is prone to upper respiratory tract obstruction such as retrolingual fall, thus increase the risk of perioperative respiratory complications. Therefore, it is very important to achieve a rapid and effective antagonistic muscle relaxant effect, reduce the postoperative muscle relaxation residue, and maintain the patency of the patient's airway.

Compared with the traditional cholinesterase inhibitor neostigmine, sugammadex is a specific antagonist of novel aminosteroid muscle blockers, which rapidly reverses moderate and deep neuromuscular block by combining with rocuronium or vecuronium 1:1,without compatibility with due to its no effect on muscarinic receptors or plasma cholinesterase. The absence of cholinergic and cardiovascular effects during awakening from anesthesia would be significant benefit for patients with cardiovascular or respiratory diseases.

The pharmacological effect of sugammadex is its ability to form a tight 1:1 complex with amino steroid neuromuscular blockers, which causes a lower plasma concentration of free neuromuscular blockers and promotes the transfer of neuromuscular blockers from the peripheral compartment (including the neuromuscular junction) to the plasma gradient. A meta-analysis by Vaghiri et al showed that reversal of neuromuscular block by sugammadex accelerated postoperative recovery of intestinal peristalsis in patients undergoing colorectal surgery compared with acetylcholinesterase inhibitors. Deljou et al confirmed that reversal of neuromuscular blockade with sugammadex shortened the time to first postoperative defecation in patients compared with neostigmine / glononium bromide. The study will investigate the effect of sugammadex in patients undergoing laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
1. Study purpose This study intends to compare the neuromuscular block effects of sugammadex or neostigmine against rocuronium after laparoscopic bariatric surgery, investigate the effect of sugammadex reversing neuromuscular block on the recovery quality of laparoscopic bariatric surgery by observing the time from muscle relaxation antagonism to TOF ratio ≥0.9, tracheal extubation time, postoperative Richmond Agitation-Sedation Scale, postoperative Visual Analogue Scale and opioid consumption, postoperative respiratory and gastrointestinal function, postoperative QoR-15 recovery quality score and other indicators, to provide clinical data for rapid recovery of laparoscopic bariatric surgery.
2. Study design

   2.1. Type of the study The research is a single-center, double-blind, randomized-controlled clinical trial.

   2.2 Sample size calculation The estimated sample size was calculated using SPSS Statistics, version 26.0 ((IBM Corp), and this was based on our preliminary study.

   2.3 Randomization and blinding

   Patients were randomly assigned in a 1:1 ratio into 2 groups, the neostigmine group or the sugammadex group via centrally computer-generated group randomization. Immediately after the surgery, a sealed opaque envelope containing the patient group assignment was opened by an experienced anesthesiologist in charge. When T2 appeared, the sugammadex group was given 2mg/kg of sugammadex intravenously (adjusted body weight), the neostigmine group was given 0.04mg/kg of neostigmine + 0.02mg/kg of atropine intravenously (adjusted body weight).

   Participants in the neostigmine group and sugammadex group were kept blinded to their group assignment. This study involved researchers who conducted the postoperative follow-up and evaluation (blinded) and researchers who administered the treatment (unblinded). The unblinded researchers who administered the interventions were not involved in the evaluation of the postoperative outcomes.
3. Quality control

   All research data, both in paper and electronic formats, will be kept for at least 5 years. If readers have any questions after the article's publication, they may contact the corresponding author for access to the original data. Patient information will remain anonymous, including name, ID number and telephone number. All data related to enrolled patients collected during the study period of this project will be archived and safeguarded, and all study members and study sponsors are asked to keep subject information confidential. The study protocol will be reviewed and revised by statistical experts. Investigators will adhere to pre-defined standard operating procedures, encompassing patient screening, follow-up standardization, result assessment, and data management. The Ethics Committee of Shanxi Bethune Hospital will review the trial every six months.
4. Statistical analysis

Statistical analysis was performed using SPSS Statistics, version 26.0. Normally distributed continuous variables were presented as mean (SD) values, and intergroup comparisons used independent-sample t-test. Nonnormally distributed variables were presented as median (IQR) values, and intergroup comparisons were determined using the Mann-Whitney test. Categorical variables were expressed as frequencies and percentages, and these were compared using either the χ2 test or the Fisher exact test. A P<0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Body Mass Index (BMI) ≥ 40kg/m²
* American Society of Anesthesiologists (ASA) grade I to III classification
* NYHA cardiac function grade I - II

Exclusion Criteria:

* Patients with neuromuscular disease or respiratory system disease
* Patients with severe abnormal liver and renal function
* Perioperative use of drugs known to interact with rocuronium
* Patients with unstable mental illness or refusal to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative muscle relaxation recovery | After injection of muscle relaxation antagonist, an average of 30 minutes
  Postoperative muscle relaxation recovery, measured using the time of train-of-four stimulation (TOF) ratio ≥0.9

SECONDARY OUTCOMES:
Postoperative pain scores at rest and during coughing | 1, 6, 12, 24 and 48 hours after surgery
  Pain scores, measured using the Visual Analog Scale(0 points indicated no pain, a score <4 indicated mild pain; a 4-7 score indicated moderate pain, a score >7 points indicated severe pain, and a score of 10 indicated unbearably severe pain)
Postoperative opioid consumption | 48 hours after surgery
  The total amount of sufentanil used in the PCA pump within the initial 48 hours postoperatively
Postoperative remedial analgesia rate | 48 hours after surgery
  The rate of remedial analgesia 48 hours postoperatively
Postoperative arterial blood gas | 12, 24 and 48 hours after surgery
  PaO2 and PaCO2, measured using the blood-gas analyzer
Postoperative pulmonary function | 12, 24 and 48 hours after surgery
  Forced expiratory volume in the first second/forced vital capacity (FEV1/FVC) and interstitial forced expiratory flow 25%-75%(FEF25%-75%) are measured using the pulmonary function testing equipment.
Postoperative gastrointestinal function | 12, 24 and 48 hours after surgery
  I-FEED scores(an I-FEED scores of 0-2 indicates postoperative gastrointestinal normality, 3-5 indicates postoperative gastrointestinal intolerance, and ≥6 indicates postoperative gastrointestinal dysfunction)
The time of first exhaust and defecation | 48 hours after surgery
  The time of first flatus and defecation within 48h after operation was measured by hour
Postoperative recovery quality | 24 and 48 hours after suegery
  Quality of recovery, measured using the 15-item Quality of Recovery questionnaire (QoR-15), It ranges from 0 to 150, with a higher score indicating a better quality of recovery

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Wen Zhang, MD, Principal Investigator — Shanxi Bethune Hospital